CLINICAL TRIAL: NCT01381055
Title: Double-blind Placebo Controlled Trial Using Pentoxifylline Associated With Pentavalent Antimony in Cutaneous Leishmaniasis
Brief Title: Antimony Plus Pentoxifylline in Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Paulo Roberto Lima Machado (Other)
Collaborators: Instituto Nacional de Ciência e Tecnologia de Doenças Tropicais (INCT-DT) (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Federal University of Bahia (Other)
Responsible Party: Sponsor-Investigator, Paulo Roberto Lima Machado, Associate Researcher, Hospital Universitário Professor Edgard Santos
Organization: Hospital Universitário Professor Edgard Santos (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCPX2011
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous leishmaniasis; Pentoxifylline; Meglumine antimoniate; L. braziliensis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline plus antimony (Experimental)
  Interventions: Drug: Pentoxifylline
- Placebo plus antimony (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Patients with cutaneous leishmaniasis treated with pentavalent antimony/Meglumine antimoniate 20mg/kg/day during 20 days and pentoxifylline pills 400mg three times a day during 20 days.
  Arms: Pentoxifylline plus antimony
Drug: Placebo — Patients with cutaneous leishmaniasis treated with pentavalent antimony/metilglucamine 20mg/kg/day during 20 days and placebo pills three times a day during 20 days.
  Arms: Placebo plus antimony

SUMMARY:
The purpose of this study is to determine whether pentoxifylline associated to pentavalent antimony has a higher cure rate than pentavalent antimony alone in the treatment of cutaneous leishmaniasis.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (untreated) cutaneous leishmaniasis with localized lesions and a positive culture or diagnosed by polymerase chain reaction (PCR) methods or by intradermal skin testing (Montenegro test).
* Number of lesions: 1 to 3 ulcerative lesions.
* Lesion´s diameter: 1 to 5 cm.
* Disease duration: up to three months.

Exclusion Criteria:

* Safety concerns:

  * AST, ALT >3 times upper limit of normal range
  * Serum creatinine or BUN >1.5 times upper limit of normal range
  * Evidence of serious underlying disease (cardiac, renal, hepatic or pulmonary)
  * Immunodeficiency or antibody to HIV
  * Any non-compensated or uncontrolled condition, such as active tuberculosis, malignant disease, severe malaria, HIV, or other major infectious diseases
  * Lactation, pregnancy (to be determined by adequate test) or inadequate contraception in females of childbearing potential for treatment period plus 2 months
* Lack of suitability for the trial:

  * Negative parasitology (aspirate/biopsy/PCR)or negative Montenegro test
  * Any history of prior anti-leishmania therapy
  * Any condition which compromises ability to comply with the study procedures
* Administrative reasons:

  * Lack of ability or willingness to give informed consent (patient and/or parent / legal representative)
  * Anticipated non-availability for study visits/procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cure rate or complete cicatrization of the ulcer. | 6 months
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.
  Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.

SECONDARY OUTCOMES:
Initial cure rate or complete cicatrization of the ulcer | 2 months
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.
  Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Roberto L Machado, MD, PhD, Principal Investigator — Federal University of Bahia
Locations (1):
- Posto de Saúde de Corte de Pedra, Corte de Pedra, Tancredo Neves/Bahia, Brazil